CLINICAL TRIAL: NCT03679000
Title: Periconceptional Phthalates Exposure and Its Epigenetic Effect on Fertility, Embryo Development, and Neonatal Outcomes: a Prospective Study
Brief Title: The Effect of Periconceptional Phthalates Exposure on Couples' Reproductive Health
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Liyufeng, Principal Investigator, Tongji Hospital
Other Study IDs: H0425
Record Dates: First submitted 2018-09-10; First posted 2018-09-20 (Actual); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Environmental Exposure; Infertility
Keywords: environmental exposure; epigenetic process; embryo development; infertility; cohort study
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Urine,serum, blastocyst culture medium for both spouse. Sperm for men. Follicular fluid for women.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- The reproductive health of couples: The study is a prospective cohort study, and its participants are childbearing couples who are seeking assisted reproductive technologies for having a baby in the reproductive center in Tongji Hospital.The study is a observational study.

SUMMARY:
The study is a prospective cohort study, which is aiming to explore periconceptional phthalates exposure and its potential epigenetic effect on fertility, embryo development, and neonatal outcomes.

DETAILED DESCRIPTION:
The study is a prospective cohort study, and its subjects are childbearing couples who are seeking assisted reproductive technologies for having a baby in the reproductive center in Tongji Hospital.

1. All enrolled couples will be needed to sign an informed consent and complete a questionnaire for collecting information about demographics, life-style, and medical and reproductive histories.
2. Biological samples will be collected from the participants to measure phthalates metabolites in order to evaluate the exposure of single person or the couple in different time phase.The samples include urine, blood that will be left after the hormones measurement for both spouses. The follicular fluid will be obtained from females on the day of oocyte retrieval. The left sperm samples after sperm analysis will be obtained from men. In the reproductive center of Tongji Hospital, hormone measurement for women and sperm analysis for men are required for the In vitro fertilization and embryo transfer in order to evaluate the fertility of couples.And the blastocyst culture medium will be obtained from couples after blastocyst transfer. All samples will be stored at -80℃ until further analysis.
3. Measurements of phthalates metabolites in the biological samples.
4. Collecting data from electronic medical records and follow-up.The basic information, clinical data and reproductive outcomes of the subjects will be collected by reviewing the electronic medical charts, including the height, weight, basic hormone levels, stimulation protocol and time, insemination protocol, fertilization rate, cleavage rate, excellent embryo rate, blastocyst formation rate, clinical pregnancy rate, as well as live birth rate，the newborns' height, weight, and gestational age, etc.
5. Analyze the miRNA expression profiles of blastocyst culture medium.
6. Statistical analysis. The investigators will analyze the association between the couples' phthalates exposure levels and the reproductive outcomes, and explore the association among periconceptional phthalates exposure, epigenetic changes and reproductive outcomes.

ELIGIBILITY:
一. Inclusion and exclusion criteria for primary study:

The exclusion of men:

1. Occupational exposures
2. Couples living in separate places
3. Congenital diseases

   * Congenital azoospermia
   * Ejaculation dysfunction
   * Family history of genetic diseases
4. Acquired diseases

   * Genitourinary infections
   * Mumps
   * Endocrine diseases
   * Sexually transmitted diseases
   * Hyperthyroidism
   * Liver failure
   * Renal failure
   * Neurological diseases
   * Paraplegia
   * Acquired testicular injury
5. Patient who have received surgeries：

   * Inguinal hernia surgery
   * Vasectomy
   * Bladder neck surgery
   * Pelvic surgery
6. Patients who have used antitumor drugs and hormone

The exclusion of women:

1. Occupational exposures
2. Couples living in separate places
3. Congenital gonadal dysplasia

   * Genital malformation
   * Chromosomal abnormalities
   * Family history of genetic diseases
4. Endocrine and metabolic diseases

   * Diabetes
   * Hyperprolactinemia
   * Thyroid and adrenal diseases
5. Cardiovascular diseases

   * Dyslipidemia
   * Systemic lupus erythematosus
   * Other rheumatic immune diseases
6. Patients who have received the following treatment:

   * Ovarian surgery
   * Thyroid surgery
   * Pituitary surgery
   * Anti-tumor radiotherapy
   * Chemotherapy
7. Patients with previous history as followed:

   * Endometrial injury
   * Endometrial polyps
   * Endometritis
   * Uterine fibroids
   * Endometriosis
8. Tubal effusion

二. Inclusive and exclusive criteria for blastocyst culture medium collection at the later stage.

Inclusion criteria:

1. Subjects in the primary part of the study
2. ·Normal gender of men and women

   * No genetic diseases or congenital diseases
   * No family genetic history
3. Normal sperm analysis for men
4. Female age <35 years
5. ·Normal Ovarian function for women

   * Normal endocrine function for women
   * No uterine disease or abnormality
6. The causes of infertility :

   * Tubal factors
   * Unexplained
7. The protocol of controlled ovary hyperstimulation :

   * A routine long-term protocol

Exclusion criteria:

1. Subjects with smoking or alcohol abuse in the past 3 months
2. Patients with overweight or obesity (BMI ≥ 25)
3. Embryos with chromosomal abnormalities confirmed by PGS

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is a group of childbearing couples who are seeking assisted reproductive technologies for having a baby in the reproductive center in Tongji Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 2122 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Phthalates exposure levels | 12/2021
  Concentrations of phthalates in ng/ml

SECONDARY OUTCOMES:
Exposure characteristics of phthalates | 12/2021
  The exposure of different personal care products in weeks
Reproductive outcomes | 12/2021
  The different reproductive outcomes in percent
The expression profiles of miRNA | 12/2021
  The expression profiles of miRNA in different quantity

CONTACTS AND LOCATIONS:
Overall Officials: Yufeng Li, Doctor, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
The reason that we do not plan to share IPD is that each participant enrolled in our study wil signed an informed consent.In the informed consent, we pledged that all information of participants will be kept strictly confidential.

REFERENCES:
- [Background] Du YY, Fang YL, Wang YX, Zeng Q, Guo N, Zhao H, Li YF. Follicular fluid and urinary concentrations of phthalate metabolites among infertile women and associations with in vitro fertilization parameters. Reprod Toxicol. 2016 Jun;61:142-50. doi: 10.1016/j.reprotox.2016.04.005. Epub 2016 Apr 8. PMID 27067915
- [Background] Wang YX, Zeng Q, Sun Y, You L, Wang P, Li M, Yang P, Li J, Huang Z, Wang C, Li S, Dan Y, Li YF, Lu WQ. Phthalate exposure in association with serum hormone levels, sperm DNA damage and spermatozoa apoptosis: A cross-sectional study in China. Environ Res. 2016 Oct;150:557-565. doi: 10.1016/j.envres.2015.11.023. Epub 2015 Dec 3. PMID 26654563
- [Background] Wang YX, You L, Zeng Q, Sun Y, Huang YH, Wang C, Wang P, Cao WC, Yang P, Li YF, Lu WQ. Phthalate exposure and human semen quality: Results from an infertility clinic in China. Environ Res. 2015 Oct;142:1-9. doi: 10.1016/j.envres.2015.06.010. Epub 2015 Jun 15. PMID 26087406
- [Background] Zeng Q, Chen YZ, Xu L, Chen HX, Luo Y, Li M, Yue J, Liu AL, Li YF, Lu WQ. Evaluation of exposure to trihalomethanes in tap water and semen quality: a prospective study in Wuhan, China. Reprod Toxicol. 2014 Jul;46:56-63. doi: 10.1016/j.reprotox.2014.03.005. Epub 2014 Mar 13. PMID 24632126
- [Background] Zeng Q, Li M, Xie SH, Gu LJ, Yue J, Cao WC, Zheng D, Liu AL, Li YF, Lu WQ. Baseline blood trihalomethanes, semen parameters and serum total testosterone: a cross-sectional study in China. Environ Int. 2013 Apr;54:134-40. doi: 10.1016/j.envint.2013.01.016. Epub 2013 Feb 26. PMID 23454109